CLINICAL TRIAL: NCT01895712
Title: Safety and Performance Registry for an All-comers Patient Population With the Limus Eluting Orsiro Stent System Within Daily Clinical Practice - III Canada
Brief Title: BIOFLOW-III Israel Satellite Registry
Status: Completed | Type: Observational
Sponsor: BIOTRONIK Israel (Industry)
Responsible Party: Sponsor
Other Study IDs: G1227
Record Dates: First submitted 2013-07-05; First posted 2013-07-10 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Diabetes Mellitus Type 1 or 2
Keywords: International; Multicenter; Observational registry; Orsiro Drug Eluting Stents (DES); Stenting; Treatment of Coronary Artery Disease; Coronary revascularization; Percutaneous Coronary Intervention (PCI); Diabetes Mellitus Type 1; Diabetes Mellitus Type 2; STEMI; NSTEMI; Ischemia; Angina; Subgroups; Acute Myocardial Infarction; Small vessels; Chronic Total Occlusion
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Ischemia; Angina Pectoris

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Orsiro

SUMMARY:
BIOTRONIK - SaFety and Performance Registry for a diabetic patient population with the .bimus Eluting Orsiro Stent System Within daily clinical practice - III

DETAILED DESCRIPTION:
For the majority of Coronary Artery Disease (CAD), treatment with Percutaneous Transluminal Coronary Angioplasty (PTCA) provides high initial procedural success. However, the medium to long-term complications range from rather immediate elastic recoil or vessel contraction to longer processes like smooth muscle cell proliferation and excessive production of extra cellular matrix, thrombus formation and atherosclerotic changes like restenosis or angiographic re-narrowing. The reported incidence of restenosis after PTCA ranges from 30%-50%. Such rates of recurrence have serious economic consequences. Bare Metal Stents (BMS), designed to address the limitations of PTCA, reduced the angiographic and clinical restenosis rates in de novo lesions compared to PTCA alone and decreased the need for CABG. BMS substantially reduced the incidence of abrupt artery closure, but restenosis still occurred in about 20%-40% of cases, necessitating repeat procedures. The invention of Drug Eluting Stents (DES) significantly improved on the principle of BMS by adding an antiproliferative drug (directly immobilized on the stent surface or released from a polymer matrix), which inhibits neointimal hyperplasia. The introduction of DES greatly reduced the incidence of restenosis and resulted in a better safety profile as compared to BMS with systemic drug administration. These advantages and a lower cost compared to surgical interventions has made DES an attractive option to treat coronary artery disease.

An interesting group of analysis resulted to be diabetic patients. It has been concluded that the incidence of both nonocclusive and occlusive restenosis is higher in diabetic subjects after stenting as judged from comparison with historical control subjects. Results implicate accelerated restenosis as both a consequence of diabetes and a cause for increased mortality after PCI in diabetic patient.

Therefore this observational registry has been designed for the clinical evaluation of the Orsiro LESS in diabetic subjects (Diabetic patients type 1 or 2) requiring coronary revascularization with Drug Eluting Stents (DES). Results will contribute to the collection of clinical evidence for the clinical performance and safety of the Orsiro Drug Eluting Stent System in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus Type 1 or 2
* Stable coronary patients with moderate-severe symptomatic angina (CCS ≥II) and evidence of myocardial ischemia per non- invasive test (nuclear or echo) or patients with 'silent' myocardial ischemia and a large (e.g. >10% of myocardium) territory of myocardium in jeopardy (nuclear or echo)
* Subject signed informed consent
* Subject is geographically stable and willing to participate at all follow up assessments
* Subject is ≥ 18 years of age

Exclusion Criteria:

* Subject did not sign informed consent
* Left main disease
* Complex bifurcations
* Ostial lesions
* Three vessel disease
* Large visible thrombus
* Heavy calcified lesions needing atherectomy or cutting balloon dilatation
* Syntax Score ≥33
* Active bleeding
* Sepsis
* Chronic total Occlusion
* Bleeding tendency obviate dual anti platelet (DAP) intake for one year
* Hb<11/Plts,100.000/WBC<4000 or >11.00
* Pregnant or nursing subjects and those who plan pregnancy in the period up to 3 years following index procedure. (Female subjects of child- bearing potential must have a negative pregnancy test done within 28 days prior to the index procedure and contraception must be used during participation in this trial)
* Known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, antiplatelet medication specified for use in the study (clopidogrel and prasugrel and ticlopidine, inclusive), sirolimus, poly (L-lactide) poly (DL-lactide), cobalt, chromium, nickel, tungsten, acrylic and fluoro polymers or contrast sensitivity that cannot be adequately pre-medicated. Planned surgery within 6 months of PCI unless dual antiplatelet therapy will be maintained
* Currently participating in another study and primary endpoint is not reached yet.
* Other medical illness (e.g, cancer or congestive heart failure) or Known history of substance abuse (alcohol, cocaine, heroin etc.) as per physician judgment that may cause non-compliance with the protocol or confound the data interpretation or is associated with a limited life expectancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic subjects (Diabetic patients type 1 or 2) requiring coronary revascularization with Drug Eluting Stents (DES).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Target Vessel Failure (TVF) | 12 months
  Composite of cardiac death, any target vessel myocardial Infarction, coronary artery bypass graft and clinically driven target vessel revascularization)

SECONDARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months
  Composite of cardiac death, target vessel Q-wave or non-Q wave Myocardial Infarction (MI), emergent Coronary Artery Bypass Graft (CABG), clinically driven Target Lesion Revascularization (TLR)
Total death | 12 months
  Total death
Cardiac death | 12-month
  Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death I death of unknown cause and all procedurerelated deaths, including those related to concomitant treatment.
Stent Thrombosis | 12-month
  Definite/probable-ARC define
Target vessel myocardial infarction | 12-month
  Myocardial infarction will be adjudicated according to the Joint ESC/ACCF/AHA/WHF Task Force universal definition of myocardial infarction12
  • 14and on the basis of the 2010 ARC extended historical definition of myocardial infarction.
Target lesion revascularization (TLR) | 12 months
  Defined as any repeat revascularization of the target lesion

CONTACTS AND LOCATIONS:
Overall Officials: Ran Kornowski, Prof, Principal Investigator — Rabin Medical Center
Locations (6):
- Israel (6):
  - Rambam medical Center, Haifa
  - Carmel medical Center, Haifa
  - Hadassah medical Center, Jerusalem
  - Meir medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Sheba medical Center, Tel Litwinsky